CLINICAL TRIAL: NCT01198054
Title: PILOT STUDY PHASE II, Multicenter, Non-randomized, TO ASSESS THE EFFICACY AND SAFETY OF LENALIDOMIDE IN INDUCTION AND POST-INDUCTION IN PATIENTS WITH NOVO Acute Myeloid Leukemia (AML) WITH Cytogenetic Abnormality Monosomy 5
Brief Title: LENA-LMA-5:Lenalidomide in Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LENA-LMA-5
Record Dates: First submitted 2010-07-29; First posted 2010-09-09 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: AML
Keywords: AML; Lenalidomide
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomine (Experimental): Post-induction lenalidomide in patients with de novo AML with deletion 5q cytogenetic abnormality (del (5q)) or monosomy 5 (-5)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Initial dose of oral lenalidomide is 10 mg/day for 28 days every 28 days, during 6 months.
  In case of response on day 169, patient will follow a treatment extension phase. The dose of lenalidomide should be the same as the last dose for initial phase, until 24 months or progression disease

SUMMARY:
The purpose of this study is to evaluate the effectiveness of post-induction lenalidomide in patients with de novo AML with deletion 5q cytogenetic abnormality (del (5q)) or monosomy 5 (-5), who obtained complete remission after conventional induction chemotherapy. So, too, for those who no obtained response treatment (total resistance) or partial remission.

At the same time, the study evaluate the security of lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

1. Confirm the diagnosis of AML according to WHO criteria (Annex 4).
2. AML de novo (ie, patients without documented history of previous treatment with antineoplastic agents for radiotherapy or other oncological diseases, hematological or immunological, related to the development of secondary LMAs and secondary AML patients without primary MDS with del (5q) or -5 [documented history of primary MDS with transformation to LMAs]).
3. Diagnostic confirmation of the abnormality del (5q) or -5, with or without other cytogenetic abnormalities. It is not necessary that the del (5q) including band 5q31.
4. Patients who have received one cycle of induction chemotherapy consisting of a classical combination of anthracycline and cytarabine (with or without etoposide as a third agent associated), regardless of the response.
5. Patients have been evaluated the response to induction chemotherapy with anthracyclines and cytarabine (with or without etoposide as third agent partner) and were classified according to the criteria of IWG.20
6. ≤ 60 patients ineligible for allogeneic hematopoietic progenitors.
7. Patients> 60 years are not eligible for allogeneic hematopoietic stem cell, or eligible but did not have HLA-identical brother.
8. Accept the use of any contraceptive method effective in patients of childbearing age with reproductive potential (see Section 6.5 on pregnancy prevention plan).
9. Ability to understand and voluntarily sign informed consent form.
10. Age ≥ 18 years at the time of signing the informed consent form.
11. Ability and willingness to follow the schedule of study visits.

Exclusion Criteria:

1. AML secondary to treatment with cytostatic or immunosuppressive agents, myelodysplastic syndrome or other neoplastic disease.
2. AML with cytogenetic abnormalities t (15, 17), t (8; 21), t (16; 16) or inv (16) or their associated molecular rearrangements.
3. Patients who have received remission induction with a different regime to cytarabine anthracycline / - etoposide.
4. ≤ 60 patients eligible for allogeneic hematopoietic progenitors.
5. Patients> 60 years eligible for allogeneic hematopoietic stem cell transplant and who have HLA-identical brother.
6. Patients who have not been evaluated the response to induction chemotherapy (complete remission, partial remission or resistance (see Table 6).
7. ECOG 3-4.
8. Any of the following laboratory abnormalities Serum creatinine> 2.0 mg / dl (177 mmol / l). serum aspartate aminotransferase (AST) / glutamic oxalacetic transaminase serum (SGOT) or alanine aminotransferase (ALT) / serum glutamate pyruvate transaminase (SGPT)> 5.0 x upper limit of normal (ULN).

   total serum bilirubin> 3 mg / dl.
9. Patient with known positive HIV serology. No HIV test is required in the process of selection.
10. Any severe psychiatric condition or disease that prevents the patient sign the informed consent form for the patient or involves an unacceptable risk should participate in the study.
11. Any serious organic disease or condition that behave for the patient if an unacceptable risk to participate in the study.
12. Previous use of cytotoxic chemotherapy agents or experimental agents (agents are not commercially available) for the treatment of AML.
13. Pregnant or breastfeeding (see Section 6.5 on pregnancy prevention plan).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Effectivity: Duration of response with lenalidomide after conventional induction chemotherapy | 12 months
  Evaluate the effectiveness of post-induction lenalidomide in patients with de novo AML with deletion 5q cytogenetic abnormality (del (5q)) or monosomy 5 (-5), who obtained complete remission after conventional induction chemotherapy. So, too, for those who no obtained reponse treatment (total resistance) or partial remission.

SECONDARY OUTCOMES:
Safety and tolerability: Type and intensity of adverse events related with lenalidomide | 1 year
  Type and intensity of adverse events related with lenalidomide

CONTACTS AND LOCATIONS:
Overall Officials: Sanz Miguel, Dr, Principal Investigator — PETHEMA Foundation
Locations (12):
- Spain (12):
  - Hospital Clínico y Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital Juan Canalejo., A Coruña
  - Hospital General de Alicante., Alicante
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital 12 de Octubre, Madrid
  - Hospital Ramón y Cajal. Madrid, Madrid
  - H. Carlos Haya, Málaga
  - Hospital Central de Asturias., Oviedo
  - Hospital Clínico Universitario de Salamanca., Salamanca
  - Hospital Universitario Virgen del Rocío., Seville
  - Hospital La Fe de Valencia, Valencia